CLINICAL TRIAL: NCT06226324
Title: fMRI Study of Early Brain Injury in Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Inner Mongolia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: AHInnerMongolia-SLE
Record Dates: First submitted 2024-01-09; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SLE with neuropsychiatric symptoms: 1. Neuropsychiatric symptoms meeting the 1999 ACR definition
  2. Ages 18-55y
  3. Female
  4. Right-handed
  5. Can cooperate with MRI and neuropsychiatric examination
  Interventions: Other: neuropsychological test
- SLE without neuropsychiatric symptoms: 1. Patients who meet the 2019 ACR diagnostic criteria for SLE
  2. Patients without neuropsychiatric symptoms
  3. Age 18-55y
  4. Female
  5. Right-handed
  6. Able to cooperate with MRI and neuropsychiatric examination
  Interventions: Other: neuropsychological test
- Healthy control group: 1. Age and gender matched the case group
  2. Right-handed
  3. No cerebrovascular, neurological or mental diseases
  4. Can cooperate with MRI and neuropsychiatric examination
  Interventions: Other: neuropsychological test

INTERVENTIONS:
Other: neuropsychological test — The subjects were evaluated for memory, cognition, mood and sleep

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease involving multiple organs and systems. The central nervous system is one of the most commonly involved parts, and the involvement of the nervous system is called neuropsychiatric lupus, which is one of the most common complications of SLE and the main cause of death. Cognitive impairment and emotional disorders are the most common neuropsychiatric symptoms, with a prevalence of up to 80%. Studies have shown that the prevalence of NPSLE is between 37% and 95%. Compared with SLE patients, the mortality rate increases by three times. Early diagnosis and treatment play an important role in improving the quality of life of patients. fMRI has the advantages of non-invasive, in vivo and high repeatability, and can detect the brain function changes of patients early before the structural changes. This study uses fMR to compare the differences in brain function changes between SLE patients and healthy controls, explore the neuroimaging mechanism of brain injury, and provide reference for the early clinical intervene.

DETAILED DESCRIPTION:
The fMRI images of 40 SLE patients with neuropsychiatric symptoms, 40 SLE patients without neuropsychiatric symptoms and 40 healthy controls matched by sex, age and education level were collected. fMRI was selected as an evaluation method to compare the differences in brain functional changes among the three groups, and to explore the specific brain regions in the imaging of early brain injury in SLE. Neurocognitive assessment was performed on all subjects, clinical data and laboratory serum markers of SLE patients were collected, and the correlation between SLE patients and specific brain regions was analyzed, and multiple regression models were constructed to provide imaging references for early clinical diagnosis and intervention in the process of NPSLE.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender matched the case group
2. Right-handed
3. No cerebrovascular, neurological or mental diseases
4. Can cooperate with MRI and neuropsychiatric examination

Exclusion Criteria:

1. Patients with serious diseases of other systems
2. Patients with diseases of central nervous system
3. Other rheumatic immune system diseases
4. Neuropsychiatric history
5. Smokers, drug users or alcoholics
6. Contraindicated MRI

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There were 80 SLE patients (40 with and without neuropsychiatric symptoms) and 40 healthy controls
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
fMRI Study of Early Brain Injury in Systemic Lupus Erythematosus | 2 years
  Early identification of specific brain areas of brain injury in lupus patients by fMRI provides objective imaging markers for early clinical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Peng fei Qiao, Study Director — The Affiliated Hospital of Inner Mongolia Medical University
Locations (1):
- Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia, China

REFERENCES:
- [Derived] Ni S, An N, Li C, Ma Y, Qiao P, Ma X. Altered structural and functional homotopic connectivity associated with cognitive changes in SLE. Lupus Sci Med. 2024 Nov 24;11(2):e001307. doi: 10.1136/lupus-2024-001307. PMID 39581701